CLINICAL TRIAL: NCT06164470
Title: Impact of Support Groups for Patients With Non-Cystic Fibrosis Bronchiectasis on Quality of Life and Exacerbations
Brief Title: Impact of Support Groups for Patients With Non-Cystic Fibrosis Bronchiectasis
Acronym: BronchConnect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-40128
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: Support Group; Patient Education
MeSH Terms: interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Support Group (Other): Non-randomized pre-post trial, in which each participant will serve as their own control. Participants will be recruited from a bronchiectasis specialty clinic.
  Interventions: Behavioral: Support Group

INTERVENTIONS:
Behavioral: Support Group — monthly virtual patient support with multidisciplinary education for 12 sessions

SUMMARY:
BronchConnect is a prospective trial to investigate the impact of support groups on health care related quality of life in those with noncystic fibrosis bronchiectasis (NCFBE). It has been well demonstrated that participation in patient support groups improves quality of life in those who suffer from interstitial lung disease and chronic obstructive pulmonary disease, but the impact is largely unknown for those who live with NCFBE, a chronic lung disease with rising prevalence with no targeted FDA-approved therapy. NCFBE causes chronic cough, dyspnea, recurrent infections, and leads to anxiety and uncertainty. This study seeks to evaluate the impact of a virtual patient support group for patients with NCFBE through questionnaires to assess change of quality of life and anxiety, and exacerbation rates through clinical assessment.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis (NCFBE) is a chronic disease of the airways characterized by progressive damage to the airways that impairs the ability to clear mucus leading to repeated cycles of inflammation and infection. The condition is associated with chronic cough, sputum production, and exacerbations requiring antibiotics and/or hospitalizations, and as such can have a significant effect on quality of life. Incidence and prevalence have been increasing in the past twenty years, with a concurrent worsening in socioeconomic burden. Chronic cough and sputum production, use of devices for airway clearance, decreased exercise tolerance, and frequent exacerbations can all lead to embarrassment and isolation. Per the European Respiratory Society (ERS) guidelines, impairment in quality of life in patients with bronchiectasis is "equivalent in terms of scores on the St George's Respiratory Questionnaire (SGRQ) to severe chronic obstructive pulmonary disease (COPD), idiopathic pulmonary fibrosis and other disabling respiratory diseases." Patient support groups are well established for those living with these other chronic pulmonary diseases, but their efficacy is not well defined for NCFBE. This is a single center prospective interventional non-randomized pre-post study to evaluate the impact of a virtual patient support group and multidisciplinary educational program for patients with NCFBE using a mixed-methods approach seeking to compare how support groups affect quality of life, anxiety, and exacerbation rates for patients living with NCFBE. Participants will complete a series of questionnaires and will undergo assessment for severity of disease, comorbidities, and exacerbations before and after attending the group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchiectasis on computed tomography (CT) chest scan
* Bronchiectasis is the primary respiratory disease as determined by a clinician

Exclusion Criteria:

* Age < 18 years old
* Cystic fibrosis
* Traction bronchiectasis in the context of pulmonary fibrosis
* Solid organ transplant recipient
* Ability to provide informed consent
* Due to constraints of this pilot study, inability to engage in a full conversation in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Baseline, 3-months, 6-months, 12-months
  The Quality of Life-Bronchiectasis (QOL-B) is a validated questionnaire that assesses bronchiectasis symptoms and their effect on quality of life. QOL-B V3.1 is 37 items in 8 scales that each are scored 0 to 100, including respiratory symptoms, functioning, health perception, vitality, and treatment burden. We will track change for each domain over time.
Anxiety | Baseline, 3-months, 6-months, 12-months
  The General Anxiety Disorder-7 is a commonly used questionnaire that assesses clinical anxiety using 7 questions over the past 14-day period. This will be tracked for score improvement (i.e. lower) over time.

SECONDARY OUTCOMES:
Exacerbation Rate | 12-months
  An exacerbation will be defined as a deterioration in three or more of the following for at least 48 hours: cough, sputum volume and/or consistency, sputum purulence, breathlessness and/or exercise tolerance, fatigue and/or malaise, hemoptysis, and a clinician determines that a change in bronchiectasis treatment is required. Assessment will include mean exacerbation per year for the prior two years, study duration, and subsequent one year.
Participation | 12-months
  Attendance to sessions will be tracked, with acceptable marked at 66% of sessions attended through the study period.
Rate of post-group survey | 12-months
  Participants will be tracked for completion of post-support group questionnaires sent at end of every meeting to assess relevance of the session, with acceptable as at least 66% of completion of surveys through the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Zha, MD/PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hester KLM, Newton J, Rapley T, De Soyza A. Patient information, education and self-management in bronchiectasis: facilitating improvements to optimise health outcomes. BMC Pulm Med. 2018 May 22;18(1):80. doi: 10.1186/s12890-018-0633-5. PMID 29788946
- [Background] Hashem F, Merritt R. Supporting patients self-managing respiratory health: a qualitative study on the impact of the Breathe Easy voluntary group network. ERJ Open Res. 2018 Feb 9;4(1):00076-2017. doi: 10.1183/23120541.00076-2017. eCollection 2018 Jan. PMID 29450201
- [Background] Alcazar B, de Lucas P, Soriano JB, Fernandez-Nistal A, Fuster A, Gonzalez-Moro JM, Arnedillo A, Sidro PG, de Los Monteros MJ. The evaluation of a remote support program on quality of life and evolution of disease in COPD patients with frequent exacerbations. BMC Pulm Med. 2016 Nov 8;16(1):140. doi: 10.1186/s12890-016-0304-3. PMID 27821164
- [Background] Athanazio RA. Bronchiectasis: moving from an orphan disease to an unpleasant socioeconomic burden. ERJ Open Res. 2021 Oct 25;7(4):00507-2021. doi: 10.1183/23120541.00507-2021. eCollection 2021 Oct. PMID 34708118